CLINICAL TRIAL: NCT05666687
Title: An Open-label, Adaptive Design Study in Healthy Male Participants to Characterize the Occupancy of NR2B Subunit Containing NMDA Receptors in the Brain Following a Single Intravenous Dose of MIJ821 Using Positron Emission Tomography (PET) With the Radioligand [11C]Me-NB1
Brief Title: An Open-label, Adaptive Design, Positron Emission Tomography Study in Healthy Male Participants to Characterize Receptor Occupancy by MIJ821 in the Brain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: CMIJ821A02111; 2022-002317-42 (EudraCT Number)
Record Dates: First submitted 2022-12-18; First posted 2022-12-28 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Major Depressive Disorder
Keywords: NR2B receptor modulator; Healthy subject; safety; pharmacokinetics receptor occupancy; PET scan; Major Depressive Disorder; adult
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: There will be 5 Cohorts
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Experimental): MIJ821, starting dose
  Interventions: Drug: MIJ821
- Cohort 2 (Experimental): MIJ821, dose will be defined based on the results of the previous cohort(s).
  Interventions: Drug: MIJ821
- Cohort 3 (Experimental): MIJ821, dose will be defined based on the results of the previous cohort(s).
  Interventions: Drug: MIJ821
- Cohort 4 (Experimental): MIJ821, dose will be defined based on the results of the previous cohort(s).
  Interventions: Drug: MIJ821
- Cohort 5 (Experimental): MIJ821, dose will be defined based on the results of the previous cohort(s).
  Interventions: Drug: MIJ821

INTERVENTIONS:
Drug: MIJ821 — MIJ821 will be administered as an i.v. infusion

SUMMARY:
The purpose of this study is to confirm binding of MIJ821 to the NR2B-containing NMDA receptors in the human brain and assess the PC-RO relationship over time using positron emission tomography (PET).

DETAILED DESCRIPTION:
This is a Phase I, open-label, adaptive design study in healthy male participants using PET imaging with the radioligand [11C]Me-NB1 to measure occupancy of the NR2B-containing NMDA receptors by MIJ821. This exploratory study will be performed at a single clinical site and a separate PET imaging site.

Up to 10 participants will be enrolled into 5 sequential cohorts. Each participant will receive a single dose of MIJ821 as an i.v. infusion. As part of the adaptive design, the dose of MIJ821 will be changed across cohorts to achieve the primary study objective in the smallest possible number of participants.

After confirming eligibility during screening, each participant will undergo a baseline PET scan. Each participant will receive a single dose of i.v. MIJ821 during the treatment period, followed by up to two post dose PET scans. Post dose safety assessments will be performed up to End of Study visit which will happen once between Day 9 and Day 15.

ELIGIBILITY:
Key Inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study
* Healthy males, aged 23 to 55 years (inclusive), and in good health as determined by past medical history, physical and neurological examination, vital signs, electrocardiogram, and laboratory tests at Screening and Baseline (whenever applicable)
* At screening and at baseline (Day -1), vital signs after 3 minutes resting (in sitting position during screening and supine position during baseline) must be within the following ranges:
* Body temperature (otic) from 35.0 °C to 37.5 °C, inclusive
* Systolic blood pressure (BP) from 90 to 139 mmHg, inclusive
* Diastolic BP from 50 to 89 mmHg, inclusive.
* Pulse rate from 50 to 90 beats per minute, inclusive
* Participants must weigh at least 50 kg to participate in the study and must have a body mass index (BMI) within the range of 18.0 to 29.9 kg/m² at screening. BMI = body weight (kg) / height2 (m2)
* Participants must be able to communicate well with the Investigator and to comply with the requirements of the entire study, including adhering to study restrictions and visit schedule

Key Exclusion criteria:

* Hypersensitivity to NMDA antagonists (MIJ821 or other compounds with similar mechanism of action, like ketamine or compounds with similar chemical structure to ketamine) or to any excipients, local anesthetics, or anticoagulants used in this study.
* Any significant illness, including infectious diseases, which has not resolved within 2 weeks prior to baseline.
* Any of the following ECG abnormalities at Screening or Baseline:
* PR interval outside 110-200 ms
* QRS duration outside 70-120 ms
* Resting heart rate in sinus rhythm outside 50-90 bpm
* QTcF > 450 ms
* Exposure to ionizing radiation as part of a research study, which, in addition to the exposure from this study, would lead to a total effective dose of more than 10 mSv in a period of one year.
* Any history of neurological disorders, including, but not limited to any of the followings:
* Any history of stroke or known cerebrovascular disorders (e.g. aneurysm or arteriovenous malformation) or known aneurysmal vascular disease in other location (e.g. aorta)
* Any history or presence of epilepsy or of seizures or convulsions of any kind.
* Any history of head trauma leading to permanent sequelae or history of head trauma leading to clinically significant but transient symptoms within 2 years of baseline.
* Score "yes" on item 4 or item 5 of the Suicidal Ideation section of the C-SSRS, if this ideation occurred in the past 6 months from screening, or "yes" on any item of the Suicidal Behavior section, except for the "Non-Suicidal Self-Injurious Behavior" (item also included in the Suicidal Behavior section), if this behavior occurred in the past 2 years.
* Sexually active males unwilling to use a condom during intercourse while taking study treatment and for 90 days following dosing. A condom is required for all sexually active male participants for 90 days following dosing (including vasectomized men) to prevent them from fathering a child AND to prevent delivery of the investigational drug via seminal fluid to their partner.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2023-01-11 (Actual); Primary Completion 2023-11-07 (Actual); Study Completion 2023-11-07 (Actual)

PRIMARY OUTCOMES:
Human Brain Receptor Occupancy and Plasma Concentration of MIJ821 | Baseline PET Scan up to 15 days post dose
  To evaluate the relationship between plasma concentration of MIJ821 and brain receptor occupancy by MIJ821 in healthy participants, by using positron emission tomography (PET) with [11C]Me-NB1

SECONDARY OUTCOMES:
Binding parameters of [11C]-MeNB1 | Baseline PET scan up to 15 days post dose
  To characterize the binding properties of [11C]-Me-NB1 in the human brain
Percentage change in PET imaging outcome measures after treatment with MIJ821 compared to baseline and plasma concentration of MIJ821 | Baseline PET scan up to 36 hours post dose
  To evaluate the relationship between displacement of central (brain) radioligand binding and systemic (plasma) concentration of MIJ821
Tmax will be calculated as a PK parameter of MIJ821 in plasma. | PK samples are collected at the end of i.v. infusion (Day 1) and at the beginning and end of each PET scan. Each cohort has 5 samples collected at various timepoints (dependent on time of PET scans) from i.v. infusion up to 5 days.
  To assess the systemic pharmacokinetics (PK) of MIJ821 after a single intravenous (i.v.) dose in healthy participants
AUC will be calculated as a PK parameter of MIJ821 in plasma | PK samples are collected at the end of i.v. infusion (Day 1) and at the beginning and end of each PET scan. Each cohort has 5 samples collected at various timepoints (dependent on time of PET scans) from i.v. infusion up to 5 days.
  To assess the systemic pharmacokinetics (PK) of MIJ821 after a single intravenous (i.v.) dose in healthy participants
Cmax will be calculated as a PK parameter of MIJ821 in plasma | PK samples are collected at the end of i.v. infusion (Day 1) and at the beginning and end of each PET scan. Each cohort has 5 samples collected at various timepoints (dependent on time of PET scans) from i.v. infusion up to 5 days.
  To assess the systemic pharmacokinetics (PK) of MIJ821 after a single intravenous (i.v.) dose in healthy participants
Number of adverse events and serious adverse events. | Baseline up to Day 15, plus 30 days
  The occurrence of adverse events must be sought by non-directive questioning of the participant at each visit during the study. Adverse events also may be detected when they are volunteered by the participant during or between visits or through physical examination findings, laboratory test findings, or other assessments (e.g., CADSS and C-SSRS).

CONTACTS AND LOCATIONS:
Overall Officials: David Steel, MD, Principal Investigator — Parexel Early Phase Clinical Unit (LONDON),
Locations (1):
- Novartis Investigative Site, Watford Road Harrow, United Kingdom

IPD SHARING:
Plan to Share IPD: No